CLINICAL TRIAL: NCT02922361
Title: Characterizing High-Cost, High-Need Patient Populations and Response to Care Management Programs at a NetworkModel Medicare Advantage Health Maintenance Organization
Brief Title: Spending and Outcomes for Complex Medicare Advantage Patients
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Amol Navathe, Principal Investigator, University of Pennsylvania
Other Study IDs: 825923
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will use data from a large network-model health maintenance organization that operates Medicare Advantage (MA) plans (CareMore) and fee-for-service Medicare data to (1) better understand the characteristics of high-need, high-cost MA enrollees patients and (2) evaluate the impact of a care management program focused on high-need high-cost MA enrollees with end-stage renal disease.

DETAILED DESCRIPTION:
There will be two aims. Aim 1 will describe and categorize high-need, high-cost populations. The investigators will use CareMore inpatient, outpatient, and pharmacy claims from years 2010-2014. The investigators will construct mortality and readmission risk category and they will utilize traditional claims-based risk models developed on out of sample data to categorize patient risk level. For the high health expenditure category, they will examine inpatient, outpatient, and pharmacy data to identify groups of patients who drive disproportionate health spending. Finally, for utilization the investigators will use claims and outpatient visit data (to the extent any electronic health record (EHR) data becomes available) to identify patients with disproportionate visit intensity. The approach to describe patients within these groups will be to categorize patients into deciles and utilize multivariate regression models to identify demographic, clinical, socioeconomic, and geographic characteristics associated with presence in a top decile along each metric. For example, the investigators will describe individual and clusters of diagnoses that are associated with high spending. They will also examine patients who meet multiple criteria and describe associated characteristics. Aim 2 will examine the impact of CareMore's end stage renal disease (ESRD) care model. They will use CareMore inpatient, outpatient, skilled nursing facilities (SNF), inpatient rehabilitation facilities (IRF), other facilities, pharmacy, and post-acute care claims and Center for Medicare and Medicaid (CMS) Fee-For-Service (FFS) data from matched geographies. They will also attempt to obtain the healthcare effectiveness data information set (HEDIS) data from health plan at patient and physician level, CMS stars measure data, available electronic medical record (EMR) data, and physician characteristics data to the extent CareMore can provide. They will perform a retrospective analysis of claims data. The investigators will use a primary comparison group of ESRD patients in Medicare FFS, particularly in localities where no ESRD special need plans (SNP) is offered to mitigate some effects of selection. The team will also explore a second comparison group of CareMore traditional MA plan enrollees who develop ESRD. They will first examine patient, physician, and plan or site characteristics associated with variation in utilization of the specialized services including enhanced nutritional counseling, personalized care plans, dialysis treatment evaluation, and supplemental medical evaluations -- using logistic regression. Second, they will perform a descriptive analysis of the association between use of these services and cost and quality outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will be patients of CareMore with at least one claim, ESRD CareMore patients enrolled in a SNP or a traditional MA plan, and Medicare FFS ESRD patients in matched geographies.

Exclusion Criteria:

* Participants without at least one claim with CareMore or not located in a matched Medicare FFS geographies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population will be all patients with at least one CareMore and CareMore ESRD patients - both enrolled in ESRD SNPs and traditional MA plan - and Medicare FFS ESRD patients in matched geographies.
Sampling Method: Non-Probability Sample
Enrollment: 61546 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months
  The study team will evaluate mortality by using 30 day mortality after readmission.

SECONDARY OUTCOMES:
Hospital Readmissions | 12 months
  The study team will evaluate re-admissions by measuring 30-day all-cause unplanned readmission.
Cost | 12 months
  The study team will evaluate cost by measuring total medical spending.
Ambulatory sensitive condition admission | 12 months
  The study team will evaluate admissions by measuring ambulatory sensitive conditions admissions.
Utilization | 12 months
  The study team will evaluate utilization be measuring the index of outpatient and inpatient utilization.

IPD SHARING:
Plan to Share IPD: No